CLINICAL TRIAL: NCT04761094
Title: Clinical Efficacy of Continuous Subcutaneous Insulin Infusion in Type 1 Diabetes Mellitus Patients in Spain
Brief Title: Clinical Efficacy of Insulin Pumps in Type 1 Diabetes Mellitus Patients in Spain
Status: Completed | Type: Observational
Sponsor: Castilla-La Mancha Health Service (Other)
Collaborators: Spanish Diabetes Association (Unknown)
Responsible Party: Principal Investigator, Jesús Moreno Fernández, Endocrinologist, Castilla-La Mancha Health Service
Other Study IDs: C-386
Record Dates: First submitted 2021-02-12; First posted 2021-02-18 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Treatment; Insulin pump; Continuous subcutaneous insulin infusion
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Infusion Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Insulin pump: All patient treated with insulin pump.
  Interventions: Device: Insulin pump

INTERVENTIONS:
Device: Insulin pump — Treatment with continuous subcutaneous insulin infusion

SUMMARY:
Observational cross-sectional multicenter study about clinical efficacy of insulin pumps in type 1 diabetes mellitus patients.

DETAILED DESCRIPTION:
Observational cross-sectional multicenter study about clinical efficacy of continuous subcutaneous insulin infusion in type 1 diabetes mellitus patients.

All clinical variables are gathered from the Spanish Insulin Pump National Registry.

Data analysis is conducted using SPSS (Chicago, IL) statistic software. Results are presented as mean +/- SD values. A paired Student's t-test or a Wilcoxon signed-rank test were used for the analysis of differences. Comparisons between proportions were analyzed using a chi-squared test. A P value < 0.05 was considered statistically significant.

The protocol was approved by the reference Castilla-La Mancha Public Health Institute Ethic Committee. All participants provided written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes patients treated with insulin pump.
* Medical treatment received in Spain.

Exclusion Criteria:

- Any other kinds of diabetes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All type 1 diabetes patients treated with continuous subcutaneous insulin infusion in Spain.
Sampling Method: Non-Probability Sample
Enrollment: 2977 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
HbA1C | During the procedure
  Glycated haemoglobin A1C

SECONDARY OUTCOMES:
TIR | During the procedure
  Time in range (TIR, 3.9-10 mmol/L, 70-180 mg/dL) of the interstitial glucose
TAR | During the procedure
  Time above range (TAR, >10 mmol/L, >180 mg/dL) of the interstitial glucose
TUR | During the procedure
  Time under range (TUR, <3.9 mmol/L, <70 mg/dL) of the interstitial glucose
Clinical significant hypoglycemia | During the procedure
  Time in clinical significant hypoglycemia (< 3 mmol/L, <54 mg/dL) of the interstitial glucose
MIG | During the procedure
  Mean interstitial glucose (mmol/L, mg/dL)
%CV | During the procedure
  Percentage of the variation coefficient (%, >36% is considered high levels)
Adherence to CGM | During the procedure
  Time of use of continuous glucose monitoring (% possible time of use)
Weight | During the procedure
  Total corporal weight (Kg)
Insulin dose | During the procedure
  Daily insulin dose requirements (UI/Kg/d)
DKA | During the procedure
  Number of diabetic ketoacidosis (number of events)
Severe hypoglycemia | During the procedure
  Number of severe hypoglycemia (number of events)
Hospital admission | During the procedure
  Number of hospital admission due to insulin pump (number of events)

CONTACTS AND LOCATIONS:
Locations (25):
- Spain (25):
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital San Joan de Deu, Esplugues de Llobregat, Barcelona
  - Hospital Universitario Mutua de Tarrasa, Terrassa, Barcelona
  - Hospital Universitario de Jerez, Jerez de la Frontera, Cadiz
  - Hospital Universitario de Santiago de Compostela, Santiago de Compostela, La Coruña
  - Hospital Infanta Sofía, San Sebastián de los Reyes, Madrid
  - Hospital Universitario Carlos Haya, Málaga, Malaga
  - Hospital Universitario Virgen de la Victoria, Málaga, Malaga
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Badajoz University Hospital, Badajoz
  - Hospital Clínic i Provincial, Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de Basurto, Bilbao
  - Obispo Rafael Torija, St., Ciudad Real
  - Centro Medico D-Medical, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid
  - Clinica DiaLibre, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Joan XXIII, Tarragona
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be available after studying each request.

REFERENCES:
- [Background] Eisenbarth GS. Type I diabetes mellitus. A chronic autoimmune disease. N Engl J Med. 1986 May 22;314(21):1360-8. doi: 10.1056/NEJM198605223142106. No abstract available. PMID 3517648
- [Background] Effect of intensive diabetes treatment on the development and progression of long-term complications in adolescents with insulin-dependent diabetes mellitus: Diabetes Control and Complications Trial. Diabetes Control and Complications Trial Research Group. J Pediatr. 1994 Aug;125(2):177-88. doi: 10.1016/s0022-3476(94)70190-3. PMID 8040759
- [Background] Yeh HC, Brown TT, Maruthur N, Ranasinghe P, Berger Z, Suh YD, Wilson LM, Haberl EB, Brick J, Bass EB, Golden SH. Comparative effectiveness and safety of methods of insulin delivery and glucose monitoring for diabetes mellitus: a systematic review and meta-analysis. Ann Intern Med. 2012 Sep 4;157(5):336-47. doi: 10.7326/0003-4819-157-5-201209040-00508. PMID 22777524
- [Background] Sastre J, Pines PJ, Moreno J, Aguirre M, Blanco B, Calderon D, Herranz S, Roa C, Lopez J; Grupo de estudio DIACAM 1. Metabolic control and treatment patterns in patients with type 1 diabetes in Castilla-La Mancha: the DIAbetes tipo 1 in Castilla La Mancha study. Endocrinol Nutr. 2012 Nov;59(9):539-46. doi: 10.1016/j.endonu.2012.07.003. Epub 2012 Oct 4. English, Spanish. PMID 23039989
- [Background] Beato-Vibora P, Chico-Ballesteros A, Gimenez M, Guerrero-Vazquez R, Barrio-Castellanos R, Goni-Iriarte MJ, Diaz-Soto G, Merino-Torres JF, Moreno-Fernandez J, Martinez-Brocca MA; Diabetes Technology Working Group of the Spanish Diabetes Association. A national survey on the efficacy and safety of continuous subcutaneous insulin infusion in patients with type 1 diabetes in Spain. Diabetes Res Clin Pract. 2018 Mar;137:56-63. doi: 10.1016/j.diabres.2017.12.009. Epub 2017 Dec 24. PMID 29278712
- [Background] Moreno-Fernandez J, Gomez FJ, Pines P, Gonzalez J, Lopez J, Lopez LM, Blanco B, Roa C, Herranz S, Munoz-Rodriguez JR. Continuous Subcutaneous Insulin Infusion in Adult Type 1 Diabetes Mellitus Patients: Results from a Public Health System. Diabetes Technol Ther. 2019 Aug;21(8):440-447. doi: 10.1089/dia.2019.0097. Epub 2019 Jun 13. PMID 31199682
- [Derived] Moreno-Fernandez J, Chico A, Martinez-Brocca MA, Beato-Vibora PI, Vidal M, Piedra M, Quiros C, Munoz-Rodriguez JR; SPAIP Registry Study. Continuous Subcutaneous Insulin Infusion in Type 1 Diabetes Mellitus Patients: Results from the Spanish National Registry. Diabetes Technol Ther. 2022 Dec;24(12):898-906. doi: 10.1089/dia.2022.0207. Epub 2022 Sep 6. PMID 35947087